CLINICAL TRIAL: NCT06275594
Title: A Prospective, Open-label, Randomized Clinical Trial to Evaluate the Efficacy and Safety of Remimazolam in patienTs Undergoing Endobronchial Ultrasound-guided Transbronchial Needle Aspiration: REST Trial
Brief Title: Trial Evaluating the Efficacy of Remimazolam in Endobronchial Ultrasound Guided Transbronchial Needle Aspiration
Acronym: REST
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, June Hong Ahn, Associate professor, Yeungnam University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YUMC2023-12-017
Record Dates: First submitted 2024-01-16; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Midazolam; Remimazolam
Keywords: Remimazolam; Midazolam; Safety; Efficacy; EBUS-TBNA
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Experimental): American Society of Anesthesiologists (ASA) I-II: initial dosing 5mg, maintenance dosing: 2.5mg, interval ≥2minutes ASA III: initial dosing 2.5mg, maintenance dosing: 1.25mg, interval ≥2minutes Remimazolam dose limitation: none Fentanyl: 25-50mcg, interval ≥5mintues, max: 200mcg
  Interventions: Drug: Byfavo
- Real world Midazolam (Active Comparator): Initial dosing 2-3mg, maintenance dosing: 0.5-1mg, interval ≥2minutes Remimazolam dose limitation: 7.5mg Fentanyl: 25-50mcg, interval ≥5mintues, max: 200mcg
  Interventions: Drug: Midazolam
- On label Midazolam (Active Comparator): <60years old and healthy: initial dosing 1.75mg, maintenance dosing: 1.0mg, interval ≥2minutes
  ≥60years old or debilitated/chronically ill: initial dosing 1.0mg, maintenance dosing: 0.5mg, interval v2minutes Remimazolam dose limitation: 7.5mg Fentanyl: 25-50mcg, interval ≥5mintues, max: 200mcg
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Byfavo — For induction and maintenance of sedation
  Other Names: Remimazolam
  Arms: Remimazolam
Drug: Midazolam — For induction and maintenance of sedation
  Arms: On label Midazolam; Real world Midazolam

SUMMARY:
Study to evaluate the efficacy and safety of remimazolam in patients undergoing endobronchial ultrasound-guided transbronchial needle aspiration

Primary Outcome Evaluate and compare the success of the procedure in patients undergoing EBUS-TBNA (Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration) when administered with remimazolam in the experimental group, versus Real world midazolam (Control Group 1), and On label midazolam (Control Group 2).

Secondary Outcome In patients undergoing EBUS-TBNA, compare the following aspects when administered with remimazolam in the experimental group versus Real world midazolam (Control Group 1) and On label midazolam (Control Group 2): Procedure start time, Time taken to achieve full alertness, Need for flumazenil administration, Total dose of fentanyl used, Scale of coughing/discomfort/convenience, Changes in vital signs, Complications related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 18 and above
2. ASA 1-3
3. BMI 18.5~30.0
4. Saturation pulse oximeter (SpO2) ≥ 90% in ambient air or with no more than 2 liters/min of O2 support
5. Patients who can comply with the procedures according to this clinical study protocol and who have voluntarily signed the consent form themselves

Exclusion Criteria:

1. Patients undergoing radial EBUS or electromagnetic navigation bronchoscopy (ENB) simultaneously
2. ASA 4 or higher
3. Mallampati score 4
4. BMI < 18.5, BMI >30.0
5. Known sensitivity to benzodiazepines, flumazenil, opioids, naloxone, or a medical condition in which these agents
6. Bronchoscopy outside the bronchoscopy unit
7. chronic kidney disease on dialysis
8. Patients with a current active acute infection or uncontrolled chronic inflammatory lung disease
9. Patients considered inappropriate for the study at the investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Procedural success during EBUS-TBNA (composite outcome) | Up to the end of the procedure (up to 1 hour)
  Success of the bronchoscopy procedure, Completion of the bronchoscopy procedure, No requirement for a rescue sedative medication, In the case of remimazolam and placebo, no requirement for more than 5 top-ups of study medication within any 15 minute period; in the case of midazolam, no requirement for more than 3 doses in any 12 minute window

SECONDARY OUTCOMES:
Time to start of procedure after administration of the first dose of study medication | Time from administration of the first dose of study medication to the start of procedure (MOAA/S ≤3) (up to 1 hour)
  Modified Observer's Assessment of Alertness and Sedation (MOAA/S)≤3 MOAA/S scores: 5 = Responds readily to name spoken in normal tone [alert], 4 =Lethargic response to name spoken in normal tone, 3 = Responds only after name is called loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Responds only after painful trapezius squeeze, 0 = Does not respond to painful trapezius squeeze.
  MOAA/S scores were assessed by the investigators.
Time taken to achieve full alertness after the procedure | Time from end of the procedure to first of three consecutive MOAA/S scores =5 (up to 1 hour)
  MOAA/S=5 MOAA/S scores: 5 = Responds readily to name spoken in normal tone [alert], 4 =Lethargic response to name spoken in normal tone, 3 = Responds only after name is called loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Responds only after painful trapezius squeeze, 0 = Does not respond to painful trapezius squeeze.
  MOAA/S scores were assessed by the investigators.
Requirement for flumazenil dosage during the procedure | From the end of procedure to discharge of bronchoscopy room (up to 1 hour)
  If MOAA/S score 5 is not reached after bronchoscopy, flumazenil will be administered. Total amount of flumazenil dosage during the procedure is measured.
  MOAA/S scores: 5 = Responds readily to name spoken in normal tone [alert], 4 =Lethargic response to name spoken in normal tone, 3 = Responds only after name is called loudly and/or repeatedly, 2 = Responds only after mild prodding or shaking, 1 = Responds only after painful trapezius squeeze, 0 = Does not respond to painful trapezius squeeze.
  MOAA/S scores were assessed by the investigators.
Total fentanyl dose | From the start of procedure to the end of procedure (up to 1 hour)
  Total amount of fentanyl during the procedure
Scale of coughing/discomfort/inconvenience | After the end of procedure (up to 1 hour)
  Coughing/discomfort/convenience visual analogue scale (Patients mark a point on a straight line corresponding to their perception of the severity of the cough, discomfort, and inconvenience. VAS ranges 0-100, with 0 representing minimal severity and 100 representing maximal severity)
Changes in blood pressure | From the start of procedure to the end of procedure (up to 1 hour)
  Changes of blood pressure (mmHg) assessed by 5 minutes
Changes of heart rate | From the start of procedure to the end of procedure (up to 1 hour)
  Changes of heart rate (rates/minutes) assessed by 5 minutes
Changes in respiration rate | From the start of procedure to the end of procedure (up to 1 hour)
  Changes of respiration rate (rates/minutes) assessed by 5 minutes
Complications related to the procedure | Up to 1 month
  Procedure related complications during 1 month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University Hospital, Daegu, Namgu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seol HY, Hong KS, Jang JG, Moon SM, Kim SH, Cho JY, Yang B, Kim S, Choi CM, Ji W, Ahn JH. A prospective, open-label, randomized clinical trial to evaluate the efficacy and safety of remimazolam in patients undergoing EBUS-TBNA: REST trial design. BMC Pulm Med. 2024 May 17;24(1):243. doi: 10.1186/s12890-024-03067-w. PMID 38760702